CLINICAL TRIAL: NCT02123381
Title: Changes in Tumor Tissue and Serum Biomarkers Before and After Cetuximab Combined With Preoperative Radiotherapy in Locally Advanced Middle or Lower Thoracic Esophageal Squamous Cell Carcinoma
Brief Title: Changes in Tumor Tissue and Serum Biomarkers Before and After Cetuximab Combined With Preoperative Radiotherapy in Locally Advanced Thoracic Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Southwest Hospital, China (Other); Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, LI TAO, Section Head, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: scch2014019
Record Dates: First submitted 2014-04-13; First posted 2014-04-25 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Locally Advanced Thoracic Middle-lower Segment Esophageal Squamous Cell Carcinoma
Keywords: tumor tissue and serum biomarkers; cetuximab; preoperative radiotherapy; esophageal squamous cell carcinoma
MeSH Terms: conditions — Neoplasms; Esophageal Squamous Cell Carcinoma | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm A (Experimental): All patients in the arm receive cetuximab combined with preoperative radiotherapy at first. 4-6 weeks after the rdiaotherapy，patients receive right thoracotomy with three incisions radical surgery.
  Interventions: Radiation: preoperative radiotherapy; Drug: cetuximab

INTERVENTIONS:
Radiation: preoperative radiotherapy — Patients receive intensity modulated radiation therapy(IMRT) or image-guided radiation therapy(IGRT)from week 1 to week 4,once a day, 5 times per week.
  Radiotherapy dose：95% gross tumor volume（GTV-T） 40Gy/20f，GTV-N 40Gy/20f，CTV-T 40Gy/20f，CTV-N 40Gy/20f.
Drug: cetuximab — 400mg/m2/week, 2 hours,iv,at week 1;250mg/m2/week,1hour,iv,at week 2-4
  Other Names: Erbitux; C225

SUMMARY:
This study aim to investigate Changes in tumor tissue and serum biomarkers before and after cetuximab combined with preoperative radiotherapy in locally advanced thoracic middle-lower segment esophageal squamous cell carcinoma.We want to find one or more effective biomarkers to predict and evaluate the patients who will be benefit from cetuximab combined with preoperative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

(1)18 to 65 years old,male or female (2)Pathologically or cytologically proven thoracic middle-lower esophageal squamous cell carcinoma; (3)clinical stage II or stage III; (4)Primary tumors can be measured; (5)Karnofsky score >70; (6)Estimated life expectancy of at least 12 weeks; (7)reproductive age women should ensure that before entering the study period contraception; (8)Hemoglobin≥90.0g/dL,white blood cell count（WBC）≥ 4000 cells/mm³,Platelet count≥100,000 cells/mm³; (9)Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal,bilirubin normal; (10)Creatinine normal OR creatinine clearance ≥ 60 mL/min; (11)Patients have good compliance to treatment and follow-up of acceptance; (12)Forced expiratory volume in one second（FEV1） ≥ 1.5 litre or ≥ 75% of the reference value; (13)Considered operable (i.e. appropriate organ functions and ability to undergo general anesthesia); (14)No severe or uncontrolled cardiovascular disease; (15)No active uncontrolled infection;

Exclusion Criteria:

1. Patient who have distant metastasis
2. The primary tumor or lymph node already received surgical treatment (except for biopsy);
3. Patient who received radiotherapy for primary tumor or lymph node;
4. Patient who received the the epidermal growth factor targeted therapy;
5. Patient who received chemotherapy or immunotherapy;
6. Patient who suffered from other malignant tumor;
7. Epidermal growth factor receptor（EGFR）mutation（-）;
8. Patient who have taken other drug test within 1 month;
9. Pregnant woman or Lactating Women and Women in productive age who refuse to take contraception in observation period;
10. Subject with a severe allergic history or idiosyncratic;
11. Subject with severe pulmonary and cardiopathic disease history; Refuse or incapable to sign the informed consent form of participating this trial;
12. Drug abuse or alcohol addicted;
13. Subject with a Personality or psychiatric diseases, people with no legal; capacity or people with limited capacity for civil conduct;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Expression of Survivin protein in Esophageal Squamous Cell Carcinoma before and after Radiotherapy | before radiotherapy and 1 months after the radiotherapy
  Survivin, an inhibitor of apoptosis protein, is highly expressed in most cancers and associated with radiotherapy resistance, increased tumor recurrence, and shorter patient survival.
Expression of p53 in Esophageal Squamous Cell Carcinoma before and after Radiotherapy | before radiotherapy and 1 months after the radiotherapy
  p53 (also known as protein 53 or tumor protein 53), is a tumor suppressor protein that in humans is encoded by the TP53 gene.p53 is important in multicellular organisms and involved in preventing cancer.
changes of serum vascular endothelial growth factor（VEGF）level before and after radiotherapy | before radiotherapy and 1 months after the radiotherapy
  Vascular endothelial growth factor (VEGF) is a signal protein produced by cells that stimulates vasculogenesis and angiogenesis.

SECONDARY OUTCOMES:
Quality of life (QOL) | up to 3 years
  Quality of life (QOL) as measured by European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30）
Overall survival | up to 3 years
  time from randomization to death
PFS（progression-free survival） | up to 3 years
  time from randomization to one of the following events, whichever comes first:
  1. Tumor progression at any time (progression of primary tumor or local lymph nodes, appearance of new lesions)
  2. Recurrence at local, regional or distant site after surgery
  3. Death from any cause
local control rate（LCR） | up to 3 years
  Time to locoregional failure after R0 resection
Pathological remission | 1 months after the end of surgery
grade 3-5 adverse events | up to 3 years
  Grade 3-5 adverse events as assessed by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0，such as esophagitis、pneumonitis and hematologic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: YONGTAO HAN, MD, PhD, Principal Investigator — Sichuan Cancer Hospital and Research Institute; GE WANG, MD, PhD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University; TAIQIAN GONG, MD, PhD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University; LONG CHEN, MD, PhD, Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University; NAIQUAN MAO, MD, PhD, Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University; ZHIHUA RUAN, MD, PhD, Principal Investigator — Southwest Hospital, China; GANG XIONG, MD, PhD, Principal Investigator — Southwest Hospital, China; JIANGUO SUN, MD, PhD, Principal Investigator — Xinqiao Hospital of Chongqing; GUANGHUI LI, MD.PHD, Principal Investigator — Xinqiao Hospital of Chongqing; DEZHI LI, MD, PhD, Principal Investigator — Xinqiao Hospital of Chongqing; MINGZHANG XIANG, MD,PhD, Principal Investigator — Xinqiao Hospital of Chongqing
Locations (1):
- Sichuan Cancer Hospital & Institute, Chengdu, Sichuan, China